CLINICAL TRIAL: NCT06715280
Title: Switching Sildenafil to Riociguat in Chronic Thromboembolic Pulmonary Hypertension After Balloon Pulmonary Angioplasty
Brief Title: Switching of Sildenafil to Riociguat in CTEPH Patients
Acronym: S2R
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, GuangMing Tan, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023.577
Record Dates: First submitted 2024-11-26; First posted 2024-12-04 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
Keywords: CTEPH; BPA; Riociguat; Sildenafil
MeSH Terms: interventions — riociguat

STUDY DESIGN:
Intervention Model Description: Prospective, open-labelled, single-arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with Chronic Thromboembolic Pulmonary Hypertension (Other): Patients with Chronic Thromboembolic Pulmonary Hypertension under Sildenafil treatment
  Interventions: Drug: Riociguat (Adempas)

INTERVENTIONS:
Drug: Riociguat (Adempas) — Oral riociguat administered according to established dose-adjustment scheme. Riociguat will be administered starting at at 1mg three times per day. If patient systolic blood pressure maintains at 95mmHg or higher, the dose will be increased 0.5mg every 2 weeks up to a maximum dose 2.5mg three times per day over 8-week period

SUMMARY:
This study was designed to investigate the safety and efficacy of replacing phosphodiesterase 5 inhibitors (PDE5i) with riociguat in patients with Chronic thromboembolic pulmonary hypertension (CTEPH) who have undergone pulmonary angioplasty (BPA) and remains symptomatic despite treatments with PDE5i.

DETAILED DESCRIPTION:
Chronic thromboembolic pulmonary hypertension (CTEPH) results from the obstruction of the pulmonary arteries by organised fibrotic thrombi and the associated microvasculopathy, leading to increased pulmonary vascular resistance and progressive right-sided heart failure. CTEPH is associated with significant mortality and morbidity, so prompt initiation of treatments are necessary to improve the prognosis.

For those with accessible pulmonary arteries occlusions, surgical pulmonary endarterectomy (PEA) is the treatment of choice. Nevertheless, about 40% of CTEPH patients are not considered to be operable due to occlusion of distal pulmonary vessels. For patients with inoperative CTEPH, current treatment options include balloon pulmonary angioplasty (BPA) and medical therapies.

Several medical therapies that target microvascular components of CTEPH, such as phosphodiesterase type 5 inhibitor (PDE5i) and endothelin receptor antagonist (ERA), have been used off-label, as the efficacy of those medications in inoperable CTEPH has not been proven in randomised controlled trials or registry data. The CHEST-1 randomised controlled trial demonstrated that the soluble guanylate cyclase stimulator (sGCs), riociguat, significantly reduced pulmonary vascular resistance and improved exercise capacity in patients with inoperative CTEPH or persistent or recurrent pulmonary hypertension after PEA. Based on the finding of this study, riociguat has been approved for treatment for symptomatic inoperable patients with CTEPH.

Both PDE5i and sGCs act via the same nitric oxide (NO)-soluble guanylate cyclase (sGC)-cyclic guanosine monophosphate (cGMP) pathway, but these two classes of medications target different molecular targets in the same pathway. PDE5i inhibits the degradation of cGMP, so its efficacy is dependent on a functioning NO-sGC-cGMP axis and the presence of intracellular cGMP. In contrast, riociguat stimulates sGC directly, thus it increases intracellular cGMP level regardless the presence of NO. Therefore, based on this biological rationale, it is postulated that riociguat may be more effective in increasing intracellular cGMP compared to PDE5i. Currently there is no head-to-head trials comparing the efficacy of PDE5i and riociguat in treating pulmonary hypertension. Nevertheless, 2 clinical trials have demonstrated improvement in the clinical and biochemical parameters after switching from PDE5i to sGCs in selected patients with pulmonary arterial hypertension (PAH) with insufficient response to PDE5i. It is currently unknown whether this switching will also apply to patients with CTEPH as those 2 clinical trials do not include patients with CTEPH.

In addition to medical therapies, BPA, an endovascular procedure to dilate the occlusions and stricture in segmental or subsegmental pulmonary arteries, has emerged as a treatment for patients with inoperable CTEPH or persistent or recurrent pulmonary hypertension after PEA. Two randomised controlled trials comparing BPA and riociguat have demonstrated that BPA was associated with a greater improvement in mean pulmonary artery pressure and reduction in pulmonary vascular resistance in inoperable CTEPH patients.

Currently, the data of safety and efficacy of switching PDE5i to sGCs after BPA is lacking. Therefore, this study was designed to investigate the safety and efficacy of replacing PDE5i with riociguat in patients with CTEPH who have undergone BPA and remains symptomatic despite treatments with PDE5i.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with established diagnosis of CTEPH who are symptomatic after Balloon pulmonary angioplasty (BPA)
2. Patients who are on stable maximally tolerated dose of sildenafil for at least 6 weeks as monotherapy, or in combination with other pulmonary hypertension specific therapies
3. WHO functional class III at screening
4. Stable dose of diuretics (if used) for at least 30 days at screening
5. No recent hospitalisation due to pulmonary hypertension or heart failure for at least 30 days

Exclusion Criteria:

1. Previous treatment with riociguat other sGCs, or documented severe drug reaction or intolerance to sGCs
2. Use of nitrates or nitric oxide donors (eg, nitroglycerin, amyl nitrite, isosorbide dinitrate etc) by any administration routes within 30 days of screening
3. Pregnant women or breast-feeding women, or women with childbearing potential not using of combination of two effective contraception methods throughout study
4. Renal impairment with glomerular filtration rate <15mL /min
5. Child-Pugh C hepatic impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2026-07-22 (Estimated); Study Completion 2027-01-22 (Estimated)

PRIMARY OUTCOMES:
Change in mean pulmonary artery pressure (mPAP) | 26 weeks
  Change in mean pulmonary artery pressure (mPAP) measured in right heart catheterization at baseline and at week 26. Pulmonary hypertension (PH) is defined as pulmonary artery pressure (PAP) ≥ 25 mmHg. And the normal resting PAP is 8-20 mmHg.
Change in pulmonary vascular resistance (PVR) | 26 weeks
  Change in pulmonary vascular resistance (PVR) measured in right heart catheterization at baseline and at week 26. Pulmonary vascular resistance (PVR) is similar to systemic vascular resistance (SVR) except it refers to the arteries that supply blood to the lungs.

SECONDARY OUTCOMES:
Change in cardiac output (CO) | 26 weeks
  Change in cardiac output (CO) measured in right heart catheterization. Cardiac output (CO) is the product of the heart rate (HR), i.e. the number of heartbeats per minute (bpm), and the stroke volume (SV), which is the volume of blood pumped from the left ventricle per beat.
Change in cardiac index (CI) | 26 weeks
  Change in cardiac index (CI) measured in right heart catheterization. The cardiac index (CI) is a hemodynamic measure that represents the cardiac output (CO) of an individual divided by their body surface area (BSA). It is crucial in assessing patients with heart failure and other cardiovascular conditions
Change in pulmonary artery wedge pressure (PAWP) | 26 weeks
  Change in pulmonary artery wedge pressure (PAWP) measured in right heart catheterization. It is the pressure measured by wedging a pulmonary artery catheter with an inflated balloon into a small pulmonary arterial branch
Change in The World Health Organization (WHO) functional class | 26 weeks
  Change in WHO functional class describes how severe a patient's pulmonary hypertension (PH) symptoms. There are four different classes - I is the mildest and IV the most severe form of PH.
Change in N-terminal pro b-type natriuretic peptide (NT-proBNP) level | 26 weeks
  Change in NT-proBNP level which is a protein that's an "ingredient" for making the BNP hormone. Like BNP, your heart makes larger amounts of NT-proBNP when it has to work harder to pump blood.
Change in walk distance by 6-minutes walk test | 26 weeks
  Change in walk distance by 6-minutes walk test which is a sub-maximal exercise test used to assess aerobic capacity and endurance.
Change in Pulmonary Embolism Quality of Life Questionnaire (PEmb-QoL) score | 26 weeks
  Change in Pulmonary Embolism Quality of Life Questionnaire score which is a reliable instrument to specifically assess Quality of Life following Pulmonary Embolism, which is helpful in the identification of patients with decreased Quality of Life following acute Pulmonary Embolism.
Change in REVEAL lite 2 risk score | 26 weeks
  Change in REVEAL lite 2 risk score which is quickly calculate patient's risk score and to help determine whether treatment escalation may be needed
Change in tricuspid regurgitation pressure gradient (TRPG) | 26 weeks
  Change in tricuspid regurgitation pressure gradient (TRPG) which reflects the difference in pressure between the right ventricle and right atrium on echocardiogram
Change in tricuspid annular plane systolic excursion (TAPSE) | 26 weeks
  Change in tricuspid annular plane systolic excursion (TAPSE) which a parameter of global RV function which describes apex-to-base shortening on echocardiogram

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Kam THH, Kam KKH, Wong MKL, Yan BPY, Tan G. Haemodynamic and clinical impacts of switching phosphodiesterase-5 inhibitors to riociguat in patients with chronic thromboembolic pulmonary hypertension (CTEPH) after balloon pulmonary angioplasty (BPA) - a prospective cohort study. BMC Pulm Med. 2026 Jan 3;26(1):42. doi: 10.1186/s12890-025-04069-y. PMID 41484960